CLINICAL TRIAL: NCT06607419
Title: Efficacy Study of Blinatumomab Clean Up Early Residual Disease for Newly Diagnosed Pediatric B Lymphoblastic Leukemia
Acronym: BBClean
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Fujian Children's Hospital (Unknown); Zhangzhou Affiliated Hospital of Fujian Medical University (Other); Guizhou Provincial People's Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); Dalian Women and Children's Medical Center (Unknown); The Third Xiangya Hospital of Central South University (Other); Hunan Provincial People's Hospital (Other); Ningbo Women & Children's Hospital (Other); Anhui Provincial Children's Hospital (Other); Jiangxi Province Children's Hospital (Other); Yuying Children's Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Shuhong Shen, Chair of hematology oncology department of SCMC, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBC-ALL2024-1
Record Dates: First submitted 2024-09-04; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: B-Cell Lymphoblastic Leukemia
Keywords: Children; B-Cell Lymphoblastic Leukemia; Blinatumomab
MeSH Terms: conditions — Burkitt Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Blinatumomab (Experimental): Patients in this group should receive Blinatumomab
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Recruited patients will receive Blinatumomab since day 29 of induction for 14 days.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of Blinatumomab in pediatric patient with newly diagnosed acute B-Lymphoblastic leukemia with poor response to early chemotherapy, i.e. day 19 MRD ≥ 0.1% (low-risk) or day 19 MRD ≥ 0.01% (intermediate-risk). The main question is:

• If the flow cytometric MRD negative (<0.01%) rate and the NGS- MRD negative (<0.0001%) rate at the end of induction for patients received Blinatumomab will be superior to historical control (D46MRD in the CCCG-ALL2020 protocol).

Participants will:

* Take 14 days full dose Blinatumomab;
* With bone marrow evaluated before and after Blinatumomab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 1 month to younger than 18 years.
* Diagnosis of acute lymphoblastic leukemia by bone marrow morphology.
* Immunophenotyping: acute B-lymphoblastic leukemia;
* Meet one of the following situations:

A. Provisional low-risk: D19MRD ≥ 0.1%; B. Provisional intermediate-risk: D19MRD ≥ 0.01%;

* Subjects in the sytudy group or their guardians must be able to understand and accept the informed consent approved by the Ethics Committee

Exclusion Criteria:

* sIgM+;
* ALL evolved from chronic myeloid leukemia (CML);
* Down's syndrome, or major congenital or hereditary disease with organ dysfunction;
* Other secondary leukemias;
* CNS involvement;
* History of epilepsy; or convulsions within the last month;
* Known underlying congenital immunodeficiency or metabolic disease;
* Congenital heart disease with cardiac insufficiency;
* Treated with glucocorticoids for ≥14 days, or ABL kinase inhibitors for > 7 days within one month before enrollment, or any chemotherapy or radiotherapy within 3 months before enrollment (except for emergency radiotherapy to relieve airway compression);
* Initial diagnosis of high risk;
* D46MRD ≥1%.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
The flow cytometric MRD | From the date of Blinatumomab completion to one week after its treatment course
  The flow cytometric MRD negative (<0.01%) rate at the end of induction for patients received Blinatumomab will superior to historical control (D46MRD in the CCCG-ALL2020 protocol)
The NGS- MRD | From the date of Blinatumomab completion to one week after its treatment course
  The NGS- MRD negative (<0.0001%) rate at the end of induction for patients received Blinatumomab will superior to historical control (D46MRD in the CCCG-ALL2020 protocol)

SECONDARY OUTCOMES:
5-year EFS | 5 years since the last recruited patient completed Blinatumomab.
  The 5-year EFS of study group was significantly higher than that of the control group.
Adverse events | From day 19 of induction therapy until the start of the second high-dose methotrexate regimen.
  Comparison of adverse events in study and control groups
Healthcare costs | Six-month since window phase
  Comparison of healthcare costs in study and control groups

OTHER OUTCOMES:
Effects of Blinatumomab on immune function | From the day of or before Blinatumomab to 3-7 days after termination of Blinatumomab.
  Immune cell subgroup, T-cell activation, depletion, and cytokine releasing will be studied before Blinatumomab and day 7 and day 14 during Blinatumomab, and 1 week after Blinatumomab discontinuation.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Anhui Provincial Children's Hospital, Hefei, Anhui
  - Fujian Children's Hospital, Fuzhou, Fujian
  - Shanghai Children's Medical center, Shanghai, Shanghai Municipality
  - Ningbo Women and Children's Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clements JD, Zhu M, Kuchimanchi M, Terminello B, Doshi S. Population Pharmacokinetics of Blinatumomab in Pediatric and Adult Patients with Hematological Malignancies. Clin Pharmacokinet. 2020 Apr;59(4):463-474. doi: 10.1007/s40262-019-00823-8. PMID 31679130
- [Background] Dreier T, Lorenczewski G, Brandl C, Hoffmann P, Syring U, Hanakam F, Kufer P, Riethmuller G, Bargou R, Baeuerle PA. Extremely potent, rapid and costimulation-independent cytotoxic T-cell response against lymphoma cells catalyzed by a single-chain bispecific antibody. Int J Cancer. 2002 Aug 20;100(6):690-7. doi: 10.1002/ijc.10557. PMID 12209608
- [Background] Gokbuget N, Dombret H, Giebel S, Bruggemann M, Doubek M, Foa R, Hoelzer D, Kim C, Martinelli G, Parovichnikova E, Maria Ribera J, Schoonen M, Tuglus C, Zugmaier G, Bassan R. Blinatumomab vs historic standard-of-care treatment for minimal residual disease in adults with B-cell precursor acute lymphoblastic leukaemia. Eur J Haematol. 2020 Apr;104(4):299-309. doi: 10.1111/ejh.13375. Epub 2020 Jan 24. PMID 31876009
- [Background] Gokbuget N, Dombret H, Bonifacio M, Reichle A, Graux C, Faul C, Diedrich H, Topp MS, Bruggemann M, Horst HA, Havelange V, Stieglmaier J, Wessels H, Haddad V, Benjamin JE, Zugmaier G, Nagorsen D, Bargou RC. Blinatumomab for minimal residual disease in adults with B-cell precursor acute lymphoblastic leukemia. Blood. 2018 Apr 5;131(14):1522-1531. doi: 10.1182/blood-2017-08-798322. Epub 2018 Jan 22. PMID 29358182
- [Background] Horibe K, Morris JD, Tuglus CA, Dos Santos C, Kalabus J, Anderson A, Goto H, Ogawa C. A phase 1b study of blinatumomab in Japanese children with relapsed/refractory B-cell precursor acute lymphoblastic leukemia. Int J Hematol. 2020 Aug;112(2):223-233. doi: 10.1007/s12185-020-02907-9. Epub 2020 Jun 20. PMID 32564243
- [Background] Kantarjian H, Stein A, Gokbuget N, Fielding AK, Schuh AC, Ribera JM, Wei A, Dombret H, Foa R, Bassan R, Arslan O, Sanz MA, Bergeron J, Demirkan F, Lech-Maranda E, Rambaldi A, Thomas X, Horst HA, Bruggemann M, Klapper W, Wood BL, Fleishman A, Nagorsen D, Holland C, Zimmerman Z, Topp MS. Blinatumomab versus Chemotherapy for Advanced Acute Lymphoblastic Leukemia. N Engl J Med. 2017 Mar 2;376(9):836-847. doi: 10.1056/NEJMoa1609783. PMID 28249141
- [Background] Kiyoi H, Morris JD, Oh I, Maeda Y, Minami H, Miyamoto T, Sakura T, Iida H, Tuglus CA, Chen Y, Dos Santos C, Kalabus J, Anderson A, Hata T, Nakashima Y, Kobayashi Y. Phase 1b/2 study of blinatumomab in Japanese adults with relapsed/refractory acute lymphoblastic leukemia. Cancer Sci. 2020 Apr;111(4):1314-1323. doi: 10.1111/cas.14322. Epub 2020 Feb 11. PMID 31971321
- [Background] Lee DW, Santomasso BD, Locke FL, Ghobadi A, Turtle CJ, Brudno JN, Maus MV, Park JH, Mead E, Pavletic S, Go WY, Eldjerou L, Gardner RA, Frey N, Curran KJ, Peggs K, Pasquini M, DiPersio JF, van den Brink MRM, Komanduri KV, Grupp SA, Neelapu SS. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol Blood Marrow Transplant. 2019 Apr;25(4):625-638. doi: 10.1016/j.bbmt.2018.12.758. Epub 2018 Dec 25. PMID 30592986
- [Background] Loffler A, Kufer P, Lutterbuse R, Zettl F, Daniel PT, Schwenkenbecher JM, Riethmuller G, Dorken B, Bargou RC. A recombinant bispecific single-chain antibody, CD19 x CD3, induces rapid and high lymphoma-directed cytotoxicity by unstimulated T lymphocytes. Blood. 2000 Mar 15;95(6):2098-103. PMID 10706880
- [Background] Ribera JM. Efficacy and safety of bispecific T-cell engager blinatumomab and the potential to improve leukemia-free survival in B-cell acute lymphoblastic leukemia. Expert Rev Hematol. 2017 Dec;10(12):1057-1067. doi: 10.1080/17474086.2017.1396890. Epub 2017 Nov 1. PMID 29082835
- [Background] von Stackelberg A, Locatelli F, Zugmaier G, Handgretinger R, Trippett TM, Rizzari C, Bader P, O'Brien MM, Brethon B, Bhojwani D, Schlegel PG, Borkhardt A, Rheingold SR, Cooper TM, Zwaan CM, Barnette P, Messina C, Michel G, DuBois SG, Hu K, Zhu M, Whitlock JA, Gore L. Phase I/Phase II Study of Blinatumomab in Pediatric Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia. J Clin Oncol. 2016 Dec 20;34(36):4381-4389. doi: 10.1200/JCO.2016.67.3301. Epub 2016 Oct 31. PMID 27998223
- [Background] Wolf E, Hofmeister R, Kufer P, Schlereth B, Baeuerle PA. BiTEs: bispecific antibody constructs with unique anti-tumor activity. Drug Discov Today. 2005 Sep 15;10(18):1237-44. doi: 10.1016/S1359-6446(05)03554-3. PMID 16213416
- [Background] Zhou H, Yin Q, Jin J, Liu T, Cai Z, Jiang B, Li D, Sun Z, Li Y, He Y, Ma L, Gao S, Hu J, He A, Du X, Liu D, Zhang X, Ke X, Zhuang J, Han Y, Wang X, Chen Y, Gordon P, Yu D, Zugmaier G, Wang J. Efficacy and safety of blinatumomab in Chinese adults with Ph-negative relapsed/refractory B-cell precursor acute lymphoblastic leukemia: A multicenter open-label single-arm China registrational study. Hematology. 2022 Dec;27(1):917-927. doi: 10.1080/16078454.2022.2111992. PMID 36000952
- [Background] Zhu M, Wu B, Brandl C, Johnson J, Wolf A, Chow A, Doshi S. Blinatumomab, a Bispecific T-cell Engager (BiTE((R))) for CD-19 Targeted Cancer Immunotherapy: Clinical Pharmacology and Its Implications. Clin Pharmacokinet. 2016 Oct;55(10):1271-1288. doi: 10.1007/s40262-016-0405-4. PMID 27209293
- [Background] Hogan LE, Brown PA, Ji L, Xu X, Devidas M, Bhatla T, Borowitz MJ, Raetz EA, Carroll A, Heerema NA, Zugmaier G, Sharon E, Bernhardt MB, Terezakis SA, Gore L, Whitlock JA, Hunger SP, Loh ML. Children's Oncology Group AALL1331: Phase III Trial of Blinatumomab in Children, Adolescents, and Young Adults With Low-Risk B-Cell ALL in First Relapse. J Clin Oncol. 2023 Sep 1;41(25):4118-4129. doi: 10.1200/JCO.22.02200. Epub 2023 May 31. PMID 37257143
- [Background] Jabbour E, Short NJ, Senapati J, Jain N, Huang X, Daver N, DiNardo CD, Pemmaraju N, Wierda W, Garcia-Manero G, Montalban Bravo G, Sasaki K, Kadia TM, Khoury J, Wang SA, Haddad FG, Jacob J, Garris R, Ravandi F, Kantarjian HM. Mini-hyper-CVD plus inotuzumab ozogamicin, with or without blinatumomab, in the subgroup of older patients with newly diagnosed Philadelphia chromosome-negative B-cell acute lymphocytic leukaemia: long-term results of an open-label phase 2 trial. Lancet Haematol. 2023 Jun;10(6):e433-e444. doi: 10.1016/S2352-3026(23)00073-X. Epub 2023 May 12. PMID 37187201
- [Background] van der Sluis IM, de Lorenzo P, Kotecha RS, Attarbaschi A, Escherich G, Nysom K, Stary J, Ferster A, Brethon B, Locatelli F, Schrappe M, Scholte-van Houtem PE, Valsecchi MG, Pieters R. Blinatumomab Added to Chemotherapy in Infant Lymphoblastic Leukemia. N Engl J Med. 2023 Apr 27;388(17):1572-1581. doi: 10.1056/NEJMoa2214171. PMID 37099340
- [Background] Chen H, Gu M, Liang J, Song H, Zhang J, Xu W, Zhao F, Shen D, Shen H, Liao C, Tang Y, Xu X. Minimal residual disease detection by next-generation sequencing of different immunoglobulin gene rearrangements in pediatric B-ALL. Nat Commun. 2023 Nov 17;14(1):7468. doi: 10.1038/s41467-023-43171-9. PMID 37978187
- [Background] Svaton M, Skotnicova A, Reznickova L, Rennerova A, Valova T, Kotrova M, van der Velden VHJ, Bruggemann M, Darzentas N, Langerak AW, Zuna J, Stary J, Trka J, Fronkova E. NGS better discriminates true MRD positivity for the risk stratification of childhood ALL treated on an MRD-based protocol. Blood. 2023 Feb 2;141(5):529-533. doi: 10.1182/blood.2022017003. PMID 36240445
- [Background] Jabbour EJ, Short NJ, Jain N, Jammal N, Jorgensen J, Wang S, Wang X, Ohanian M, Alvarado Y, Kadia T, Sasaki K, Garris R, Garcia-Manero G, Ravandi F, Kantarjian HM. Blinatumomab is associated with favorable outcomes in patients with B-cell lineage acute lymphoblastic leukemia and positive measurable residual disease at a threshold of 10-4 and higher. Am J Hematol. 2022 Sep;97(9):1135-1141. doi: 10.1002/ajh.26634. Epub 2022 Jun 24. PMID 35713551